CLINICAL TRIAL: NCT04230694
Title: Continuous Glucose Monitoring of Hospitalized Patients With Diabetes: A Pilot Study to Establish Evidence
Brief Title: Continuous Glucose Monitoring of Hospitalized Patients With Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 018-601
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-07

CONDITIONS: Diabetes; Diabetes Mellitus; Glucose, High Blood; Glucose, Low Blood
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Dexcom Generation 6 CGM (Dexcom Gen6) device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (Active Comparator): Control Group subjects will wear the CGM device during their hospitalization, up to 10 days, but glucose readings will NOT be continuously monitored. Control Group subjects will have their glucose management guided by routine standard of care finger sticks. The readings from the CGM device are recorded and reviewed retrospectively, but not used for glucose management during the hospital stay.
  Interventions: Device: Dexcom Generation 6 CGM (Dexcom Gen6) device
- Treatment Group (Experimental): Treatment Group subjects will wear the CGM device during their hospitalization, up to 10 days, and glucose readings WILL be continuously monitored. Treatment Group subjects will have their glucose management guided by readings from the CGM device and standard of care finger sticks.
  Interventions: Device: Dexcom Generation 6 CGM (Dexcom Gen6) device

INTERVENTIONS:
Device: Dexcom Generation 6 CGM (Dexcom Gen6) device — Standing orders for blood sugars less than 100 will allow for administration of glucose replacement in the intervention group based on Dexcom Gen6 readings.
  Other Names: CGM

SUMMARY:
Systematic continuous glucose monitoring (CGM) is commonly provided as a treatment option to patients with diabetes in ambulatory care settings yet is rarely provided during hospitalization. CGM of inpatients has the potential to be the care delivery innovation that is feasible, cost effective and can improve glucose control, especially by reducing hypoglycemic events. Studies of CGM use in the ICU setting have been found to be helpful for reducing hypoglycemia in some studies while less so in others, however, these studies were performed with earlier generation glucose monitoring devices(5). ICU studies have confirmed accuracy of CGM measurements compared with capillary glucose even in settings with use of vasopressors and large-volume resuscitation. A limited number of studies have evaluated glycemic outcomes in the inpatient non-ICU setting. Studies of non-ICU patients (6-10) are limited by very small sample size, short study duration, and use of older CGM devices. There is, therefore, a critical need to systematically investigate the use of CGM in the inpatient care of patients with diabetes mellitus who are receiving care in a hospital setting that is typical of inpatient care.

DETAILED DESCRIPTION:
AIM

1) Test the health impact of CGM of inpatients as defined by rates of hypo- and hyperglycemia and the derivative of time in appropriate glucose range. Forty (40) patients will be randomized 1:1 into one of two conditions. In the treatment condition, patients will receive a Dexcom Gen6 device and the clinical staff (i.e., nursing and medical staff assigned to the patient's care) will be trained to use readings from the Dexcom Gen6 for the management of the patient's glucose levels below 100. In the control condition, patients will receive a Dexcom Gen6 device, but the clinical staff (i.e., nursing and medical staff assigned to the patient's care) will not have access to the readings and will provide usual care (four glucose checks per 24 hours and use of insulin or other diabetic agent ordered by the admitting and rounding providers to determine glucose management).

1. Hypothesis 1: Patients in the treatment condition will experience fewer episodes of hypoglycemia as compared to patients in the control condition as measured by the Dexcom Gen6 readings.
2. Hypothesis 2: Patients in the treatment condition will experience less frequent hyperglycemia events as compared to patients in the control condition as measured by the Dexcom Gen6 readings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 and Type 2 diabetes.
* Subjects 18 years of age or older with diabetes.
* Subjects willing to avoid using high dose acetaminophen (defined as greater than 4 gm per day)
* Subjects with expected hospital length-of-stay of 2 or more days beyond the time of enrollment.
* Subjects willing to wear CGM device.

Exclusion Criteria:

* Female subjects who are pregnant or lactating at the time of enrollment into the study. Females with childbearing potential will be queried about the possibility of pregnancy and a serum pregnancy test will be performed.
* Subjects with greater than 4gm use of Tylenol/24 hr.
* Surgical patients or patients with pre-planned surgery or procedure in the next 48 hours.
* Subjects with acute illness admitted to the ICU or expected to require admission to the ICU.
* Patients who may potentially require IV insulin.
* Patients with skin lesions, severe psoriasis, burns, tattoos, scarring, redness, infection or edema at the application sites that could interfere with device placement or the accuracy of interstitial glucose measurements.
* Patient with a known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Patients who have had organ transplant.
* Patients with any severe medical conditions such as end-stage renal disease on dialysis, status post renal transplantation, end-stage liver disease with diffuse anasarca, heart failure on inotropic support, Ejection Fraction (EF) < 15 % or severe sepsis.
* Any condition for which, in the opinion of the investigators, it would not be in the best interest of the participant.
* Legally protected subjects (under judicial protection, guardianship, or supervision), persons deprived of their liberty, mental or language barriers rendering the subject unable to understand the nature, scope and possible consequences of the study.
* Subjects with active substance abuse.
* Subjects with infaust prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Hypoglycemia Events during hospitalization | Up to 10 days
  Dexcom Gen6 readings

SECONDARY OUTCOMES:
Number of Hyperglycemia Events during hospitalization | Up to 10 days
  Dexcom Gen6 readings

CONTACTS AND LOCATIONS:
Overall Officials: Tresa McNeal, MD, Principal Investigator — Baylor Scott & White Medical Center - Temple
Locations (1):
- Baylor Scott & White Medical Center - Temple, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Levetan CS, Passaro M, Jablonski K, Kass M, Ratner RE. Unrecognized diabetes among hospitalized patients. Diabetes Care. 1998 Feb;21(2):246-9. doi: 10.2337/diacare.21.2.246. PMID 9539990
- [Background] Mendez CE, Mok KT, Ata A, Tanenberg RJ, Calles-Escandon J, Umpierrez GE. Increased glycemic variability is independently associated with length of stay and mortality in noncritically ill hospitalized patients. Diabetes Care. 2013 Dec;36(12):4091-7. doi: 10.2337/dc12-2430. Epub 2013 Oct 29. PMID 24170754
- [Background] Curkendall SM, Natoli JL, Alexander CM, Nathanson BH, Haidar T, Dubois RW. Economic and clinical impact of inpatient diabetic hypoglycemia. Endocr Pract. 2009 May-Jun;15(4):302-12. doi: 10.4158/EP08343.OR. PMID 19502209
- [Background] Rubin DJ, Golden SH. Hypoglycemia in non-critically ill, hospitalized patients with diabetes: evaluation, prevention, and management. Hosp Pract (1995). 2013 Feb;41(1):109-16. doi: 10.3810/hp.2013.02.1016. PMID 23466973
- [Background] van Steen SC, Rijkenberg S, Limpens J, van der Voort PH, Hermanides J, DeVries JH. The Clinical Benefits and Accuracy of Continuous Glucose Monitoring Systems in Critically Ill Patients-A Systematic Scoping Review. Sensors (Basel). 2017 Jan 14;17(1):146. doi: 10.3390/s17010146. PMID 28098809
- [Background] Gomez AM, Umpierrez GE, Munoz OM, Herrera F, Rubio C, Aschner P, Buendia R. Continuous Glucose Monitoring Versus Capillary Point-of-Care Testing for Inpatient Glycemic Control in Type 2 Diabetes Patients Hospitalized in the General Ward and Treated With a Basal Bolus Insulin Regimen. J Diabetes Sci Technol. 2015 Aug 31;10(2):325-9. doi: 10.1177/1932296815602905. PMID 26330394
- [Background] Schaupp L, Donsa K, Neubauer KM, Mader JK, Aberer F, Holl B, Spat S, Augustin T, Beck P, Pieber TR, Plank J. Taking a Closer Look--Continuous Glucose Monitoring in Non-Critically Ill Hospitalized Patients with Type 2 Diabetes Mellitus Under Basal-Bolus Insulin Therapy. Diabetes Technol Ther. 2015 Sep;17(9):611-8. doi: 10.1089/dia.2014.0343. Epub 2015 Apr 30. PMID 25927357
- [Background] Levitt DL, Silver KD, Spanakis EK. Inpatient Continuous Glucose Monitoring and Glycemic Outcomes. J Diabetes Sci Technol. 2017 Sep;11(5):1028-1035. doi: 10.1177/1932296817698499. Epub 2017 Mar 14. PMID 28290224
- [Background] Levitt DL, Silver KD, Spanakis EK. Mitigating Severe Hypoglycemia by Initiating Inpatient Continuous Glucose Monitoring for Type 1 Diabetes Mellitus. J Diabetes Sci Technol. 2017 Mar;11(2):440-441. doi: 10.1177/1932296816664538. Epub 2016 Aug 20. No abstract available. PMID 27543272
- [Background] Spanakis EK, Levitt DL, Siddiqui T, Singh LG, Pinault L, Sorkin J, Umpierrez GE, Fink JC. The Effect of Continuous Glucose Monitoring in Preventing Inpatient Hypoglycemia in General Wards: The Glucose Telemetry System. J Diabetes Sci Technol. 2018 Jan;12(1):20-25. doi: 10.1177/1932296817748964. Epub 2017 Dec 13. PMID 29237288
- [Background] Bradley C, Plowright R, Stewart J, Valentine J, Witthaus E. The Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) evaluated in insulin glargine trials shows greater responsiveness to improvements than the original DTSQ. Health Qual Life Outcomes. 2007 Oct 10;5:57. doi: 10.1186/1477-7525-5-57. PMID 17927832
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226

DOCUMENTS (1):
  • Study Protocol (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04230694/Prot_001.pdf